CLINICAL TRIAL: NCT03048942
Title: A Randomised Phase II Pilot Study of 3 Weekly Cabazitaxel Versus Weekly Paclitaxel Chemotherapy in the First Line Treatment of HER2 Negative Breast Cancer
Brief Title: Pilot Study of Cabazitaxel and Paclitaxel in HER2 Negative Breast Cancer
Acronym: CONCEPT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON/2012/4234
Record Dates: First submitted 2014-10-30; First posted 2017-02-09 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-05

CONDITIONS: HER2 Negative Metastatic Breast Cancer
Keywords: Breast cancer; HER2 negative; Cabazitaxel; Paclitaxel; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — cabazitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabazitaxel (Experimental): 6 cycles of cabazitaxel intravenous chemotherapy 25mg/m2 on day 1 of each 21 day cycle
  Interventions: Drug: Cabazitaxel
- Paclitaxel (Active Comparator): 6 cycles of Paclitaxel intravenous chemotherapy 80mg/m2 on days 1,8 and 15 of each 21 day cycle.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Cabazitaxel — 3 weekly cyctotoxic chemotherapy
  Other Names: Jevtana
  Arms: Cabazitaxel
Drug: Paclitaxel — Weekly cyctotoxic chemotherapy
  Arms: Paclitaxel

SUMMARY:
90 patients with HER2 negative breast cancer will be randomised to receive 18 weeks of chemotherapy treatment, either 6 cycles of 3 weekly Cabazitaxel or 6 cycles of weekly Paclitaxel to determine the difference in progression free survival between the 2 groups. If results at that stage suggest a potential benefit then the trial will be developed further to accrue 70 more patients.

DETAILED DESCRIPTION:
This is a prospective multicentre, randomised, open label, study comparing the efficacy and the safety of six 3-weekly cycles cabazitaxel versus 18 x weekly paclitaxel given as first line chemotherapy treatment in patients with HER2-normal metastatic breast cancer. Randomisation will be conducted by a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Metastatic breast cancer fit to receive cytotoxic chemotherapy for metastatic disease
* Measurable disease as per RECIST 1.1
* HER2 negative defined as ICH 0+, 1+ or 2+ and FISH/SISH/CISH(ration<2.0) in the case of IHC 2+
* ECOG performance status 0 or 1
* ER+ve or ER-ve
* Female age ≥18 years
* Anticipated life expectancy > 6 months
* Haemoglobin >10.0g/DL
* Absolute neutrophil count>1.5 x 10^9/L
* Platelet count>100 x 10^9/L
* ALT/SGPT<1.5 X ULN
* Serum creatinine <1.5 x ULN
* Negative pregnancy test for all women of child bearing potential

Exclusion Criteria:

* Grade ≥2 oral mucositis or peripheral or sensory neuropathy
* History of other malignancy
* History of severe hypersensitivity ≥grade 3 to polysorbate 80- containing drugs and taxanes
* Clinically significant cardiovascular disease
* Any acute or chronic medical condition
* Acute infection requiring systemic antibiotics or antifungal medication
* Sex hormones
* Administration of any live vaccine within 8 weeks
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5
* Participation in another clinical trial with an investigational drug within 30 days of randomisation
* Pregnant or breast feeding women
* Contraindications to the use of corticosteroid treatment
* HER2 Positive breast cancer
* Previous Paclitaxel chemotherapy in the adjuvant setting
* Previous cytotoxic chemotherapy for metastatic disease
* Palliative radiotherapy for metastatic disease within 4 weeks of randomisation
* Symptomatic brain metastases confirmed with CT/MRI brain
* History of other malignancy
* Grade 2

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-11; Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Defined as the time from randomisation to either disease progression or death from any cause, whichever came first, assessed up to 5 years.
  Duration of progression free survival

SECONDARY OUTCOMES:
Clinical benefit rate | At the completion of 6 cycles of chemotherapy, which is after 18 weeks
  Defined as stable disease rate + partial response rate+complete response rate according to RECIST 1.1 criteria
Objective response rate | At completion of 6 cycles of chemotherapy, which is after 18 weeks.
  Defined as complete and partial response recorded from the start of treatment to completion of 6 cycles of treatment.
Overall survival | Determined as the time from randomisation to death from any cause. Average survival rates for this population may be approximately 18 months.
  Survival duration from randomisation to date of death.
Time to next chemotherapy treatment | Measured from from the date of the last day of trial treatment. approximately after progression which on average would be after 12 months.
  time from randomisation to another chemotherapy treatment after confirmed progression.
Time to response | Determined by time from randomisation to radiological partial response, usually within the 6 cycles of treatment, therefore wihtin 18 weeks.
  Time taken for tumour burden to respond to treatment
Quality of life as measured by patients themselves | EQ5D-5L and FACT B will be completed at baseline, prior to cycles 3 and 5 and at the end of treatment visit, therefore within approximately 21 weeks from randomisation
  2 Quality of life questionnaires
Number of adverse events and Number of participants with adverse events per arm and the grade of AEs | Form the date of consent to 30 days after trial treatment has stopped.
  CTCAE Version 4.0 graded AEs

CONTACTS AND LOCATIONS:
Overall Officials: Amit K Bahl, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust
Locations (13):
- United Kingdom (13):
  - Imperial Healthcare NHS Trust, London, Avon
  - Royal United Hospital, Bath
  - Blackpool Victoria Hospital, Blackpool
  - Bristol Haematology and Oncology Centre, Horfield Road, Bristol
  - Velindre Cancer Centre, Cardiff
  - Royal Devon and Exeter Hospital, Exeter
  - Guy's Hospital, London
  - Freeman Hospital, Newcastle
  - City Hospital, Nottingham, Nottingham
  - Derriford Hospital, Plymouth
  - Musgrove Park Hospital, Taunton
  - Royal Cornwall and Treliske, Truro
  - Worcestershire Acute Hospitals NHS Trust, Worcester

IPD SHARING:
Plan to Share IPD: No